CLINICAL TRIAL: NCT03336840
Title: Effect of Metformin and Probiotics in Reproductive-aged Patients With Polycystic Ovary Syndrome: a Randomized, Parallel Study
Brief Title: Effect of Metformin and Probiotics in Reproductive-aged Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS2017
Record Dates: First submitted 2017-11-02; First posted 2017-11-08 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin (Experimental)
  Interventions: Drug: Metformin tablets
- Probiotics (Experimental)
  Interventions: Drug: ProMetS probiotics powder
- Metformin and Probiotics (Experimental)
  Interventions: Drug: 1. Metformin tablets; 2. ProMetS probiotics powder

INTERVENTIONS:
Drug: Metformin tablets — 0.5g (1 pill) of Metformin tablets administered three times a day orally before meal
  Arms: Metformin
Drug: ProMetS probiotics powder — 4g (2 strips) of ProMetS probiotics powder administered orally every night
  Arms: Probiotics
Drug: 1. Metformin tablets; 2. ProMetS probiotics powder — 1. 0.5g (1 pill) of Metformin tablets administered three times a day orally before meal;
  2. 4g (2 strips) of ProMetS probiotics powder administered orally every night
  Arms: Metformin and Probiotics

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness on the clinical and biological parameters of reproductive-aged PCOS women after a 12-week metformin and/or probiotics administration.

DETAILED DESCRIPTION:
Probiotics are live bacteria that offer a health benefit to the host when administered in adequate amounts. Probiotic supplementation is safe for use and has demonstrated beneficial effects for metabolic diseases such as obesity and diabetes. In this study, about 90 reproductive-aged women with PCOS will be enrolled. Participants will be randomly assigned into one of the following three groups: Metformin tablets (0.5g tid po), ProMetS probiotics powder (4g qN po), Metformin tablets (0.5g tid po) and ProMetS probiotics powder (4g qN po), for 12 weeks. Blood and stool samples will be collected before and after treatment. Fasting glucose levels, fasting insulin levels, sex hormone levels, serum lipid profiles, inflammation markers, other metabolic related parameters and change of gut microbiota and immune cells will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal between 18-40 years of age.
2. Diagnosed PCOS defined as 2003 Rotterdam diagnostic criteria.

Exclusion Criteria:

1. During the pregnancy and lactation period.
2. Significant impaired liver function, impaired renal function, mental disease, severe infection, severe anemia, severe heart disease and neutropenia disease.
3. Use of antibiotics within 3 months.
4. Symptoms of any infection at screening.
5. Immunodeficient or use of immunosuppressive drugs.
6. Use of products containing prebiotics or probiotics within the last 3 months.
7. Previous history of gastrointestinal surgery or disease (such as peptic ulcer, irritable bowel syndrome, inflammatory bowel disease or other gastrointestinal disorder).
8. Medical conditions or diseases that may affect subject safety or confound study results in the opinion of the investigator

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in menstrual cycle | 12 weeks
  Patients will be required to maintain a menstrual calendar and record their basal body temperature for the duration of the study and asked to fill a questionnaire before and after study. The questionnaire will cover menstrual cycle dates, duration and amount.
Improvement in hirsutism | 12 weeks
  Modified Ferriman and Gallwey score (m-FG scores) will be measured before and after study. M-FG score > 8 is considered hirsutism and when the score is higher, the symptom is more serious.
Improvement in acne score | 12 weeks
  Visual assessment of acne using "mild/moderate/severe" grades will be assessed before and after study.

SECONDARY OUTCOMES:
Gut microbiota | 12 weeks
Fasting glucose levels | 12 weeks
Fasting insulin levels | 12 weeks
Serum follicle-stimulating hormone levels | 12 weeks
Serum luteinizing hormone levels | 12 weeks
Serum estradiol levels | 12 weeks
Serum testosterone levels | 12 weeks
Serum lipid profiles | 12 weeks
  including triglycerides (mmol/L), total cholesterol (mmol/L), low density lipoprotein cholesterol (mmol/L), and high density lipoprotein cholesterol (mmol/L)
Inflammation markers | 12 weeks
  including C-reactive protein (mg/L)
Immune cells | 12 weeks
  including count and frequency of T-cell subpopulations like T-regulatory (Treg) cells (/ml), T-helper (Th) cells (/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China